CLINICAL TRIAL: NCT00592579
Title: Phase 2, Open-Label, Safety, and Efficacy Study of 2-Methoxyestradiol Administered to Patients With Plateau Phase or Relapsed Multiple Myeloma
Brief Title: A Phase 2 Study With Panzem in Patients With Relapsed or Plateau Phase Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Carolyn Sidor, MD, MBA; Chief Medical Officer, EntreMed, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-CL-004
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Relapsed Multiple Myeloma; Plateau Phase Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — 2-Methoxyestradiol

ARMS (1):
- 1 (Experimental): Open label, oral administration of 2ME2
  Interventions: Drug: 2-methoxyestradiol

INTERVENTIONS:
Drug: 2-methoxyestradiol — 800 mg of 2ME2 (capsules) administered orally every 12 hours for a total daily dose of 1600 mg.
  Other Names: Panzem

SUMMARY:
The purpose of the study is to determine the safety and effectiveness of providing 2-methoxyestradiol to patients with plateau phase or relapsed multiple myeloma. Information regarding trough 2ME2 levels will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Have plateau phase (patients who have been previously treated with at least one conventional or high-dose chemotherapy who are currently off all therapy for at least 4 weeks and are considered to have stable disease) or relapsed MM. Patients in plateau phase must have M-protein concentrations that are stable for at least 4 weeks prior to registration.
2. Be at least 18 years of age.
3. Have monoclonal plasma cells in the marrow.
4. have M-protein greater than or equal to 1g/dL in the serum or 200 mg of monoclonal light chain in a 24-hour urine protein electrophoresis.
5. Have laboratory data as specified below:

   * AST and ALT < 2.5 x upper limit of normal (ULN)
   * Alk phos < 5.0 x ULN
   * direct bilirubin < 2 x ULN
   * Creatinine < 3.0 x ULN
   * ANC greater than or equal to 750 cells/mm3
   * Platelets > 25,000/mm3
   * Hemoglobin greater than or equal to 7.0g/dL
6. Have life expectancy of at least 3 months
7. Have ECOG performance status of 0, 1, or 2
8. Women and men of child bearing potential must agree to use effective barrier contraceptive methods during study.
9. Have the ability to understand the reuirements of the study, provide written informed consent, abide to study restrictions, and agree to return for the required assessments.

Exclusion Criteria:

1. Be pregnant or nursing.
2. Have any condition that is likely to detrimentally affect regular follow up.
3. Have a history of myocardial infarction within the last 3 months, angina pectoris/angina equivalent in the last 3 months, or uncontrolled congestive heart failure.
4. Have an active infection
5. Have had major surgery within 21 days of starting 2ME2 administration
6. Have additional uncontrolled serious medical or psychiatric illness
7. have had any active cancer in addition to the MM within the last 5 years (excluding superficial skin cancer)
8. Have uncontrolled or untreated active bleeding or thrombotic disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2001-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To determine tumor response of 2ME2 administered orally by evaluation of objective responses in patients with plateau phase or relapsed multiple myeloma | At least yearly

SECONDARY OUTCOMES:
To assess the safety and tolerability of 2ME2 administered orally by evaluation of the frequency, severity, and duration of treatment-emergent adverse events in patients with plateau phase or relapsed multiple myeloma | As reported
To determine the minimum 2ME2 levels achieved in plasma following daily oral administration in patients with plateau phase or relapsed multiple myeloma | At least yearly

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Result] Rajkumar SV, Richardson PG, Lacy MQ, Dispenzieri A, Greipp PR, Witzig TE, Schlossman R, Sidor CF, Anderson KC, Gertz MA. Novel therapy with 2-methoxyestradiol for the treatment of relapsed and plateau phase multiple myeloma. Clin Cancer Res. 2007 Oct 15;13(20):6162-7. doi: 10.1158/1078-0432.CCR-07-0807. PMID 17947482